CLINICAL TRIAL: NCT06227988
Title: ASSESSMENT OF SURGICAL RISK IN PATIENTS WITH CHRONIC LIVER DISEASE USING VOCAL PENN SCORE
Acronym: vocal penn 01
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Other Study IDs: Vocal penn score 01
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: CHRONIC LIVER DISEASE
Keywords: Fluid buildup in the belly (ascites); Gallstones.; Muscle loss.
MeSH Terms: conditions — Ascites; Gallstones; Muscular Atrophy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with liver disease who undergoing surgery: For each patient and surgery, we will be collecting detailed pre-operative data regarding demographics (age, sex, body mass index, surgery category, comorbidities (diabetes mellitus, hypertension), and pertinent laboratory values (sodium, creatinine, total bilirubin, the international normalized ratio [INR], albumin, platelet count.) The etiology of liver disease will be classified.
  To ensure that laboratory data accurately reflected the pre-operative state, only those from within 30 days prior to surgery will be considered For each patient VOCAL PENN score, MELD score, and Mayo score will be calculated using an online calculator.
  Interventions: Procedure: patients with liver disease who undergoing surgery; Procedure: patients with liver disease who do not undergoing surgery
- patients with liver disease who do not undergoing surgery: For each patient and surgery, we will be collecting detailed pre-operative data regarding demographics (age, sex, body mass index, surgery category, comorbidities (diabetes mellitus, hypertension), and pertinent laboratory values (sodium, creatinine, total bilirubin, the international normalized ratio [INR], albumin, platelet count.) The etiology of liver disease will be classified.
  To ensure that laboratory data accurately reflected the pre-operative state, only those from within 30 days prior to surgery will be considered For each patient VOCAL PENN score, MELD score, and Mayo score will be calculated using an online calculator.
  Interventions: Procedure: patients with liver disease who undergoing surgery; Procedure: patients with liver disease who do not undergoing surgery

INTERVENTIONS:
Procedure: patients with liver disease who undergoing surgery — For each patient and surgery, we will be collecting detailed pre-operative data regarding demographics (age, sex, body mass index, surgery category, comorbidities (diabetes mellitus, hypertension), and pertinent laboratory values (sodium, creatinine, total bilirubin, the international normalized ratio [INR], albumin, platelet count.) The etiology of liver disease will be classified.
  To ensure that laboratory data accurately reflected the pre-operative state, only those from within 30 days prior to surgery will be considered For each patient VOCAL PENN score, MELD score, and Mayo score will be calculated using an online calculator.
Procedure: patients with liver disease who do not undergoing surgery — For each patient and surgery, we will be collecting detailed pre-operative data regarding demographics (age, sex, body mass index, surgery category, comorbidities (diabetes mellitus, hypertension), and pertinent laboratory values (sodium, creatinine, total bilirubin, the international normalized ratio [INR], albumin, platelet count.) The etiology of liver disease will be classified.
  To ensure that laboratory data accurately reflected the pre-operative state, only those from within 30 days prior to surgery will be considered For each patient VOCAL PENN score, MELD score, and Mayo score will be calculated using an online calculator.

SUMMARY:
4a. Primary To assess postoperative mortality at 30 and 90 days using the VOCAL PENN score

4b. Secondary To assess potential differences in prediction accuracy between VOCAL-Penn and MELD for 30 and 90-day mortality

DETAILED DESCRIPTION:
For each patient and surgery,we will be collecting detailed pre-operative data regarding demographics (age, sex, body mass index, surgery category, comorbidities (diabetes mellitus, hypertension), and pertinent laboratory values (sodium, creatinine, total bilirubin, the international normalized ratio [INR], albumin, platelet count.) The etiology of liver disease will be classified.

To ensure that laboratory data accurately reflected the pre-operative state, only those from within 30 days prior to surgery will be considered For each patient VOCAL PENN score, MELD score, and Mayo score will be calculated using an online calculator.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established cirrhosis Patients who had not received liver transplantation and who underwent surgery of interest were included These surgery categories will be the same as those used in the original VOCAL-Penn derivation study and will include the open abdominal, laparoscopic abdominal, and abdominal wall.

Exclusion Criteria:

* Patients with insufficient pre-operative data to compute the VOCAL-Penn score, Mayo risk score, or MELD-Na score will be excluded.

Patients undergoing liver surgeries Patients who received multiple surgeries Those who didn't give consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. STUDY POPULATION Data of 53 patients with liver disease who undergoing surgery of interest will be included
  2. DESIGN AND DURATION OF THE STUDY
  Prospective observational study Duration 2 years
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
To assess postoperative mortality at 30 and 90 days using the VOCAL PENN score | 2 years
  . For comparison between prediction scores receiver operative curves will be used.

SECONDARY OUTCOMES:
To assess potential differences in prediction accuracy between VOCAL-Penn and MELD for 30 and 90-day mortality | 2 years
  For subgroup analysis comparison between groups independent sample T test will be used.
  used.

CONTACTS AND LOCATIONS:
Overall Officials: PRACHITI Gokhe, Principal Investigator — AIG HOSPITALS
Locations (1):
- Dr Prachiti Gokhe, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No